CLINICAL TRIAL: NCT06959719
Title: Air Entrainment vs. Standard Treatment in Non-Expandable Lung With Persistent Pleural Effusion: A Randomised Controlled Double-Blind Trial
Brief Title: ARMSTRONG - Air entRainMent vS sTandard tReatment in nOn-expandable luNG
Acronym: ARMSTRONG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A097090
Record Dates: First submitted 2025-04-08; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Non-expandable Lung; Trapped Lung; Pleural Effusion; Malignant Pleural Effusions (Mpe)
Keywords: air entrainment; trapped lung; non-expandable lung (NEL); pleural effusion; malignant pleural effusion
MeSH Terms: conditions — Pleural Effusion; Pleural Effusion, Malignant; Myeloproliferative Disorder, Chronic, with Eosinophilia

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group, randomized controlled trial with a 2:1 allocation ratio (intervention:control). The unequal allocation was chosen to maximise the number of participants receiving the potentially beneficial intervention, following favourable initial data from service evaluation. Randomization will be performed centrally, and both participants and outcome assessors will be blinded to group allocation to minimize bias.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard practice (No Intervention): Fluid drainage will be performed according to standard practice, with cessation of fluid removal at the first sign of patient discomfort to prevent pain.
- Air Entrainment (Experimental): During pleural effusion drainage, atmospheric air will be intentionally introduced into the pleural space by opening the 3-way tap to air. This aims to reduce excessive negative pressure, which can create a vacuum effect within the pleural space and is thought to contribute to patient pain during drainage. The tap allows controlled air entry without fluid leakage, helping to minimise pain while maintaining safe drainage.
  Interventions: Procedure: Air Entrainment - intentional introduction of the atmospheric air into the pleural space.

INTERVENTIONS:
Procedure: Air Entrainment - intentional introduction of the atmospheric air into the pleural space. — This intervention is distinct in that it uses a standard 3-way tap, already present in routine pleural drainage procedures, to intentionally introduce atmospheric air into the pleural space in a controlled and repeatable manner. Unlike other studies where air entrainment may occur incidentally or as part of more invasive procedures, this method specifically utilises precise manipulation of the tap handle to allow intermittent air entry, aiming to reduce negative intrapleural pressure and associated pain during fluid drainage. Air entry is carefully controlled, can be repeated up to five times per procedure, and does not interfere with fluid drainage or introduce additional equipment or complexity.
  Arms: Air Entrainment

SUMMARY:
This is a randomised controlled trial evaluating whether controlled air introduction into pleural space (air entrainment) during pleural effusion drainage reduces pain, improves patient satisfaction, and facilitates more effective drainage in patients with non-expandable lung (NEL).

NEL lung is a common complication in patients with malignant or chronic pleural effusions, where the lung fails to fully re-expand after fluid removal due to pleural disease or fibrosis. In these patients, drainage often creates excessive negative pressure within the pleural cavity, leading to pain, vasovagal episodes, early termination of drainage, and the need for repeated procedures.

This study investigates a simple, safe, and low-cost intervention using a standard 3-way tap attached to the drainage system. By intermittently opening the tap to atmospheric air during drainage, air enters the pleural cavity in a controlled fashion, reducing negative pressure and potentially reducing pain, improving drainage tolerance, and minimising the need for repeated procedures.

Pleural effusion drainage is a common procedure in patients with advanced malignancy or chronic pleural disease. In patients with NEL, fluid removal creates a vacuum effect within the pleural space due to the inability of the lung to fully re-expand. This negative pressure is a key driver of severe procedural pain, vasovagal symptoms, and premature cessation of drainage. It may also necessitate multiple drainage procedures over a short period.

Currently, there are limited strategies to mitigate this problem, often relying on stopping the procedure prematurely or on analgesia, which does not address the underlying cause.

This trial evaluates the introduction of atmospheric air into the pleural space during drainage as a pragmatic, low-cost solution. The technique uses standard equipment - a 3-way tap - allowing air to be introduced safely and intermittently during drainage to reduce the vacuum effect.

Patients undergoing therapeutic pleural drainage with an indwelling catheter or chest drain will be randomised in a 2:1 ratio to:

Standard drainage care (control group)

Drainage with intermittent controlled air introduction (intervention group)

Air entrainment will be performed by briefly opening the 3-way tap to atmospheric air during drainage up to five times, based on patient discomfort and operator discretion. This aims to equalise pleural pressures, reduce pain, and improve drainage outcomes.

Randomisation is weighted 2:1 towards the intervention group to maximise the number of patients who may benefit, following favourable preliminary data. Both patients and outcome assessors will be blinded to group allocation.

Outcomes collected

Primary Outcomes:

Patient-reported pain scores during drainage - Pain will be assessed using the Visual Analogue Scale (VAS), ranging from 0 to 10 cm, where 0 indicates "no pain" and 10 indicates "worst imaginable pain." Higher scores represent a worse outcome.

Secondary Outcomes:

Volume of pleural fluid drained Number of pleural drainage procedures required Time interval between drainage procedures Incidence of complications (e.g., pneumothorax, re-expansion pulmonary oedema, infection) Reasons for incomplete drainage, including the presence and characteristics of non-expandable lung Patient-reported satisfaction with the drainage procedure

DETAILED DESCRIPTION:
Background and Rationale Air entrainment during pleural effusion drainage may improve pain control, increase fluid removal, and reduce repeat procedures in patients with non-expandable lung (NEL). A local evaluation showed greater pain relief than opioids without adverse events. This study compares air entrainment with standard drainage in NEL.

Objectives

Primary: Determine if air entrainment offers superior pain relief vs standard drainage.

Secondary: Compare fluid volume drained, time to repeat drainage, complication rates (infection, hypotension, air leaks, persistent pain), and patient satisfaction. The questionnaire assessed patient experience across four areas: pre-procedure, during the procedure, post-procedure, and overall care. Each item used 5-point Likert scales. Pre-procedure: Satisfaction with information, understanding, scheduling, and communication. During: Comfort, pain management, staff professionalism, and privacy. Post-procedure: Clarity of aftercare, symptom control, and follow-up. Overall: General satisfaction and likelihood to recommend.

Study Design Prospective, double-blind, randomised intervention study (2:1 ratio) at Cambridge University Hospital. All patients undergoing thoracentesis will be screened; only those with confirmed NEL will be analysed.

Randomisation Patients will be randomised 2:1 (intervention:control) to maximise exposure to the intervention. Allocation is blinded to both patients and VAS assessors.

Population

Inclusion: Adults (≥18) with suspected/confirmed NEL and persistent pleural effusion undergoing thoracentesis; English-speaking and able to consent.

Exclusion: Prior pleurodesis, active infection, baseline VAS ≥5, IPC requirement, contraindications, or inability to consent.

Sample Size 41 NEL patients (27 intervention, 14 control), allowing for 30% dropout. Powered for a 3.4 cm VAS difference (SD 3.1), power = 0.8, alpha = 0.05. Interim analysis after enrolment of 7 control and 14 intervention patients.

Interventions

Intervention: Air introduced into pleural space via 3-way tap to relieve negative pressure (up to five times/session).

Control: Standard thoracentesis, stopped at first discomfort.

Outcomes

Primary Outcome: Pain will be measured using the Visual Analogue Scale (VAS) at four time points: pre-procedure, during the procedure, immediately post-procedure, and 10-15 minutes after the procedure. The VAS is a 10 cm horizontal line with two anchors: 0 represents "no pain" and 10 represents "worst imaginable pain." Patients will be asked to mark the point on the line that corresponds to their pain level, and the distance from the 0 point will be recorded in centimeters to quantify pain intensity.

Secondary Outcomes:

Volume Drained: The total volume of fluid drained will be measured in milliliters (mL).

Time to Repeat Procedure: The time to repeat the procedure, if required, will be recorded in days.

Complications: The occurrence of complications, such as infection, hypotension, air leaks, or persistent pain, will be documented.

Satisfaction: Patient satisfaction will be assessed through a questionnaire, which evaluates various aspects of their experience, including pre-procedure communication, comfort during the procedure, pain management, post-procedure care, and overall experience. Satisfaction will be measured on a Likert scale ranging from "very satisfied" to "very dissatisfied."

Methodology Baseline VAS and clinical data collected. Procedure performed as per allocation. Post-procedure data includes VAS, fluid volume, complications, satisfaction, and follow-up for up to 6 months or until IPC/VATS/death.

Analysis Pain: t-test or Mann-Whitney U, depending on data distribution. Secondary outcomes: t-test, Mann-Whitney U, Chi-square or Fisher's exact depending on data type and distribution.

Analysis will follow the intention-to-treat (ITT) principle, with all patients analysed in their originally assigned groups. Missing data will be addressed using appropriate imputation methods (e.g., multiple imputation), and sensitivity analyses will be conducted to assess the robustness of findings under different missing data assumptions.

Ethics REC Ref: 25/LO/0128 | IRAS ID: 348247 Written informed consent required. Risks: Discomfort, minor complications. Benefits: Possible better pain control and fewer procedures.

Data Management Data stored securely in EPIC with restricted access. Consent forms digitised. Analysis based on anonymised data.

Patient and Public Involvement (PPI) Patient feedback informed the design of patient-facing study materials.

Dissemination Results will be published, presented, shared with stakeholders, and posted on the CUH website. Trial to be registered on ClinicalTrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older with a suspected or confirmed diagnosis of NEL and persistent pleural effusion.
* Patients who are scheduled for pleural effusion drainage as part of their standard care.
* Ability to adequately understand verbal or written information in English and provide informed consent in English.

Exclusion Criteria:

* Patients with a history of pleurodesis or other procedures that may affect pleural dynamics.
* Patients with active infections or other acute medical conditions that could interfere with the study.
* Patient with multifactorial pain and high baseline score pain defined as VAS >= 5
* Patients requiring IPC
* Individuals with known contraindications to pleural drainage or air entrainment.
* Patients who cannot provide informed consent in English, do not adequately understand verbal or written information in English or have special communication needs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Pain Relief | From the procedure start until 15 minutes after the procedure
  Pain will be measured using the Visual Analog Scale (VAS) before, during, and immediately after the drainage procedure and again 10-15 minutes later to capture the progression of relief.

SECONDARY OUTCOMES:
Drainage Volumes | Up to 6 months post-randomization
  The total volume of fluid removed during each drainage procedure.
Number of pleural drainage procedures required. | Up to 6 months post-randomization
  Total number of pleural drainage procedures performed during the study period.
Time interval between drainage procedures. | Up to 6 months post-randomization
  Time interval between consecutive pleural drainage procedures, measured in days, throughout the study period.
Complications | Up to 6 months post-randomization
  Incidence of procedure-related complications, including infections, hypotension, air leaks, and persistent pain.
Patient Satisfaction | At each in-person visit, through study completion (6 months)
  Assessed through a post-procedure survey using a standardised satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that may be shared includes pain scores recorded during the procedure, the volume of pleural effusion drained, any complications occurring during or after the procedure, and details of incomplete drainage, including evidence of and reasons for trapped lung. This data may be shared to support further research conducted by both commercial and non-commercial organisations, within the UK and internationally.
Supporting Information: ICF